CLINICAL TRIAL: NCT01415765
Title: Phase I/II Study of MLN4924 Alone Followed by Dose-Adjusted EPOCH-Rituximab + MLN4924 With Gene Expression Profiling and Mutational Analysis in Relapsed/Refractory de Novo Diffuse Large B-Cell Lymphoma
Brief Title: MLN4924 Compared With MLN4924 Plus Chemotherapy for Large B-cell Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110216; 11-C-0216
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-01-07

CONDITIONS: Lymphoma, Diffuse Large-Cell B-cell; Diffuse, Large B-cell Lymphoma; Lymphoma, Diffuse Large-Cell; Large-Cell Lymphoma, Diffuse
Keywords: Germinal Center Like B-Cell (GCB) DLBCL; Activated B-Cell Like (ABC) DLBCL; NF-KappaB Pathway; Drug Resistance; Nedd-8 Activating Enzyme Inhibitor; Diffuse Large B-Cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Acromesomelic dysplasia, Maroteaux type; Lymphoma | interventions — pevonedistat; Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Rituximab; Filgrastim

INTERVENTIONS:
Drug: MLN4924 — Part A: 150mg/m2 IV (in the vein) on days 1,4,7,11 of each 21 day cycle Part B: variable dose levels IV on days 1,5 each 21 day cycle
Drug: Etoposide — CIV(continuous intravenous infusion) on days 1-4 of every 21 day cycle
Drug: Prednisone — PO (by mouth) twice daily on days 1-5 of every 21 day cycle
Drug: Vincristine — CIV on days 1-4 of every 21 day cycle
Drug: Cyclophosphamide — IV on day 5 of each 21 day cycle
Drug: Doxorubicin — CIV on days 1-4 of each 21 day cycle
Drug: Rituximab — IV on day 1 of each 21 day cycle
Drug: Filgrastim — Subcutaneously beginning Day 6 of each 21 day cycle

SUMMARY:
Background:

- MLN4924 is an experimental cancer drug. It may help kill lymphoma cells and make them more sensitive to chemotherapy. EPOCH R is a combination chemotherapy drug. It has been effective in treating some cases of large B-cell lymphoma. This research will look at two things. The first is the effect of MLN4924 on its own in treating large B-cell lymphoma. The second is the safe dose and effect of MLN4924 and EPOCH-R in combination when treating large B-cell lymphoma.

Objectives:

* To study how MLN4924 affects large B-cell lymphoma tumors.
* To compare the effects of MLN 4924 alone and MLN4924 plus standard EPOCH-R chemotherapy.

Eligibility:

- Individuals at least 18 years of age who have large B-cell lymphoma that will be treated with chemotherapy.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine tests, tumor samples, and imaging studies.
* Participants will receive MLN4924 for a maximum of six 21-day cycles of treatment. Each cycle involves a dose of MLN4924 twice a week for 2 weeks, followed by a 1-week rest period. Participants will be monitored with frequent blood tests and imaging studies.
* Participants who do not benefit from MLN4924 alone will have MLN4924 along with EPOCH-R chemotherapy for up to six cycles of treatment.

DETAILED DESCRIPTION:
Background:

* Diffuse large B-cell lymphomas (DLBCL) have been molecularly sub-classified into germinal center like B-cell (GCB) and activated B-cell like (ABC) DLBCL.
* Clinically, the ABC subtype has a significantly higher rate of drug resistance and lower survival. The ABC subtype has constitutive activation of the NF-KappaB pathway which may account for the drug resistance.
* The ability of NF-KappaB to inhibit responses to cancer therapeutic agents may also contribute to the refractory clinical behavior of ABC subtype, and inhibition of NF-KappaB can synergize with chemotherapy to kill tumor cells.
* Because a phase II randomized design is not clinically or technically practical at this early stage to address the scientific endpoints, we have designed a novel endpoint based on relative efficacy of DA-EPOCH-R + MLN 4924 (DA-EPOCH-RN) in ABC and GCB DLBCL. Based on our study that shows that survival of relapsed ABC and GCB DLBCL are comparable and poor following initial R-CHOP, we hypothesize that significantly improved survival of ABC compared to GCB DLBCL after DA-EPOCH-RN is strongly indicative of preferential activity of MLN4924 in ABC DLBCL.

Objectives:

* Assess response of MLN4924 in relapsed/refractory DLBCL
* Assess toxicity and safe tolerated dose of MLN4924 and DA-EPOCH-R
* Assess difference in response (CR/PR) and OS in ABC and GCB DLBCL

Eligibility:

* Relapsed/refractory de novo DLBCL greater than or equal to 18 years.
* No PMBL DLBCL
* No patients with active CNS lymphoma.
* No pregnant or breast-feeding women.
* Adequate organ function (as defined in protocol).

Study Design:

* This is a single center with a sequential treatment design. The study is divided into two parts (A and B). Clinical end points are to assess the activity of MLN4924 alone (Part A) and in combination with DA-EPOCH-R (Part B), and to assess the toxicity and MTD of DA-EPOCH-RN.
* In Part A, MLN4924 will be given alone for 6 cycles.
* In Part B, MLN4924 will be initially escalated to determine the maximum tolerated dose (MTD) in combination with DA-EPOCH-R at dose levels (to be determined) and schedule every 21 days. Responding or stable patients may receive up to 6 cycles of DAEPOCH-RN.
* Patients will be restaged every 2 cycles during treatment, and every 3, 4 and 6 months during years one, two and three respectively, thereafter. Standard response criteria will be applied.
* A total of 56 patients will be enrolled depending on the relative differences in response observed between the ABC and GCB subtypes to MLN4924.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Biopsy-proven relapsed or refractory Large B-cell lymphoma.
* Confirmed pathological diagnosis by the Laboratory of Pathology, NCI.
* Age greater than or equal to 18 years.
* ECOG performance status 0-2.
* Adequate renal function or creatinine clearance > 50 ml/min/1.73m(2) unless lymphoma related.
* Adequate hepatic and hematological function, as defined by:

  * Bilirubin must be less than or equal to ULN, except less than or equal to 2 mg/dl (total) in patients with Gilbert s syndrome (as defined by > 80% unconjugated hyperbilirubinemia);
  * ALT and AST must be less than or equal to Grade 1.
  * ANC > 1000 and platelets > 75,000 unless lymphoma related.
  * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) must be less than or equal to 1.5 times the upper limit of the normal range (ULN); except if, in the opinion of the Investigator, the aPTT is elevated because of a positive Lupus Anticoagulant.
* Left ventricular ejection fraction (LVEF) > 45% as assessed by echocardiogram or MUGA
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patients must use an appropriate method of barrier contraception (eg, condoms), inform any sexual partners that they must also use a reliable method of contraception (ie, a hormonal contraceptive, an intrauterine device, diaphragm with spermicide, or abstinence), and refrain from blood and semen donation during the study and for 4 months after the last dose of study treatment.

EXCLUSION CRITERIA:

* Female subject pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum Beta-human chorionic gonadotropin (Beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for women without child-bearing potential.
* History of a prior invasive malignancy in past 5 year.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has greater than or equal to Grade 2 peripheral neuropathy within 14 days before enrollment
* Serious concomitant medical illnesses that would jeopardize the patient s ability to receive the regimen with reasonable safety.
* HIV positive patients
* Systemic cytotoxic therapy within 3 weeks of treatment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* CYP3A inducers within 14 days before the first dose of MLN4924. Moderate and strong CYP3A inhibitors and CYP3A inducers are not permitted during the study. Patients must have no prior history of chronic amiodarone use in the 6 months prior to the first dose of MLN4924.
* Patients currently taking statins who are unwilling or unable to refrain from using statins on the day prior to, day of, and day after each MLN4924 administration
* Diarrhea > Grade 1, based on the NCI CTCAE categorization despite use of optimal antidiarrheals
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
* Clinically uncontrolled central nervous system (CNS) involvement (Patients who have a history of CNS involvement, but no evidence of active CNS disease are not excluded.)
* Ongoing anticoagulant therapy (eg, aspirin, Coumadin, heparin) that cannot be held to permit bone marrow sampling. Patients who require anticoagulant therapy, and can not be maintained on low molecular weight heparin should not be considered for this study.

INCLUSION OF WOMEN AND MINORITIES:

-Both men and women and members of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-15; Primary Completion 2014-01-07 (Actual); Study Completion 2014-01-07 (Actual)

PRIMARY OUTCOMES:
Assess response of MLN4924 in relapsed/refractory DLBCL | 4 years
Assess toxicity and safe tolerated dose of MLN4924 and DA-EPOCH-R | 4 years
Assess ORR (CR/PR) and PFS of MLN4924 and DA-EPOCH-R in relapsed/refractory DLBCL | 4 years

SECONDARY OUTCOMES:
Analyze molecular subtype (ABC and GCB) | 4 years
Assess difference in response between ABC and GCB subtypes of relapsed/refractory DLBCL/MLN 4924 alone and w/MLN4924 and DA-EPOCH-R | 4 years
Analyze mutations of the ITAM motifs, CARD11 and A20 in DLBCL | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Rosenwald A, Wright G, Chan WC, Connors JM, Campo E, Fisher RI, Gascoyne RD, Muller-Hermelink HK, Smeland EB, Giltnane JM, Hurt EM, Zhao H, Averett L, Yang L, Wilson WH, Jaffe ES, Simon R, Klausner RD, Powell J, Duffey PL, Longo DL, Greiner TC, Weisenburger DD, Sanger WG, Dave BJ, Lynch JC, Vose J, Armitage JO, Montserrat E, Lopez-Guillermo A, Grogan TM, Miller TP, LeBlanc M, Ott G, Kvaloy S, Delabie J, Holte H, Krajci P, Stokke T, Staudt LM; Lymphoma/Leukemia Molecular Profiling Project. The use of molecular profiling to predict survival after chemotherapy for diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jun 20;346(25):1937-47. doi: 10.1056/NEJMoa012914. PMID 12075054
- [Background] Davis RE, Ngo VN, Lenz G, Tolar P, Young RM, Romesser PB, Kohlhammer H, Lamy L, Zhao H, Yang Y, Xu W, Shaffer AL, Wright G, Xiao W, Powell J, Jiang JK, Thomas CJ, Rosenwald A, Ott G, Muller-Hermelink HK, Gascoyne RD, Connors JM, Johnson NA, Rimsza LM, Campo E, Jaffe ES, Wilson WH, Delabie J, Smeland EB, Fisher RI, Braziel RM, Tubbs RR, Cook JR, Weisenburger DD, Chan WC, Pierce SK, Staudt LM. Chronic active B-cell-receptor signalling in diffuse large B-cell lymphoma. Nature. 2010 Jan 7;463(7277):88-92. doi: 10.1038/nature08638. PMID 20054396